CLINICAL TRIAL: NCT05360147
Title: Liraglutide Improve Cognitive Function in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director, Center for Hypertension and Metabolic Diseases, Department of Hypertension and Endocrinology, Daping Hospital, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LICD study
Record Dates: First submitted 2021-04-26; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Cognitive function; Liraglutide; Functional near-infrared spectroscopy; Metabolic changes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Sulfonylurea Compounds; Thiazolidinediones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): treated with oral antidiabetic drugs alone or combined with insulin, except for glucagon-like peptide type 1 (GLP-1) analogue
  Interventions: Drug: Oral antidiabetic drugs: Metformin, Sulfonylureas (2nd generation), Thiazolidinediones, α-Glucosidase inhibitors, and Glinides
- Liraglutide (Active Comparator): liraglutide started at an initial dose of 0.6 mg/day and a maximum dose of 1.8mg/day, adjusted once a week when hyperglycemia was uncontrolled
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Liraglutide is a glucagon-like peptide type 1 (GLP-1) analogue. We had fond its cognitive improvement effects in an observational study. In order to confirm the effects, the investigators conduct a randomized, controlled study.
  Arms: Liraglutide
Drug: Oral antidiabetic drugs: Metformin, Sulfonylureas (2nd generation), Thiazolidinediones, α-Glucosidase inhibitors, and Glinides — oral antidiabetic drugs (OADs) or insulin, except for glucagon-like peptide type 1 (GLP-1) analogues
  Arms: Placebo

SUMMARY:
Patients with diabetes are susceptible to dementia, but regular therapy fails to reduce the risk of dementia. In previous observational study, the investigators found that liraglutide can improve cognitive function in patients with T2DM through a metabolism-independent pathway. Here the investigators aim to further verify such effects through a randomized, controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes Mellitus

Exclusion Criteria:

* T2DM with acute diabetic complications;
* type 1 diabetes;
* other diseases affecting cognitive function (e.g., congenital dementia, brain trauma, epilepsy, severe hypoglycemic coma, cerebrovascular disease, ischemic heart disease, renal dysfunction);
* alcohol abuse, mental illness, and psychoactive substance abuse;
* history of thyroid disease;
* any surgical or medical conditions that could significantly influence the absorption, distribution, metabolism, or excretion of interventional drugs;
* unwillingness to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Changes in cognitive function from baseline to 12 weeks | 0 week, 12 week
  MMSE

SECONDARY OUTCOMES:
Changes of metabolic parameters from baseline to 12 weeks | 0 week, 12 week
  Systolic and diastolic blood pressure
Changes of Alzheimer's disease-associated serum markers from baseline to 12 weeks | 0 week, 12 week
  Aβ42
Changes of Alzheimer's disease-associated serum markers from baseline to 12 weeks | 0 week, 12 week
  tau
Changes of Alzheimer's disease-associated serum markers from baseline to 12 weeks | 0 week, 12 week
  P-tau
Changes of Alzheimer's disease-associated serum markers from baseline to 12 weeks | 0 week, 12 week
  TDP-43
Changes of Alzheimer's disease-associated serum markers from baseline to 12 weeks | 0 week, 12 week
  IL-6
Changes of Alzheimer's disease-associated serum markers from baseline to 12 weeks | 0 week, 12 week
  IL-8
Changes of Alzheimer's disease-associated serum markers from baseline to 12 weeks | 0 week, 12 week
  TNF-a
Changes of metabolic parameters from baseline to 12 weeks | 0 week, 12 week
  HbA1c
Changes of metabolic parameters from baseline to 12 weeks | 0 week, 12 week
  fasting plasma glucose
Changes of metabolic parameters from baseline to 12 weeks | 0 week, 12 week
  body mass index
Changes of metabolic parameters from baseline to 12 weeks | 0 week, 12 week
  lipid profile
Changes of metabolic parameters from baseline to 12 weeks | 0 week, 12 week
  waist circumference

CONTACTS AND LOCATIONS:
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, Chongqing Municipality, China